CLINICAL TRIAL: NCT05193695
Title: Heat or Excesice in Treadmill as Techique to Reduce Dry Needling Pain in Treatment of Trigger Points of Muscle Triceps Sural in Ankle Post Fracture Patients
Brief Title: How to Reduce Dry Needling Pain in Treatment of Trigger Points of Muscle Triceps Sural in Ankle Post Fracture Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: full sample size
Sponsor: Becerra, Pablo (Other)
Responsible Party: Principal Investigator, Pablo Yañez Becerra, Physical therapist, Becerra, Pablo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Becerra
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Physical Therapy Modalities; Pain Measurement; Trigger Point Pain, Myofascial; Ankle Fractures; Rehabilitation; Needles
Keywords: Humans; Excercise therapy; Hot temperature; Post dry needling; Range of motion, articular; Muscle Strength
MeSH Terms: conditions — Myofascial Pain Syndromes; Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Patients remained in the supine position for 20 minutes lying on a stretcher after dry needling.
- Treadmill (Experimental): The patients walked on a treadmill for 20 minutes after dry needling, with an inclination of 5 degrees and at a speed at which the perceived exertion was 5 according to the Borg CR10 scale (Chen et al., 2002).
  Interventions: Other: Treadmill exercise

INTERVENTIONS:
Other: Treadmill exercise — the patients walked on a treadmill for 20 minutes after dry needling, with an inclination of 5 degrees and at a speed at which the perceived exertion was 5 according to the Borg CR10 scale (Chen et al., 2002)
  Other Names: Treadmill after dry needling
  Arms: Treadmill

SUMMARY:
Ankle fractures are one of the main causes of hospitalization due to injuries in Chile, which also have a discharge and partial load time of approximately 12 weeks in the recovery process. This generates disuse and atrophy of the posterior musculature of the leg called the triceps sural, which makes it difficult to restart and perform the gait. We conducted this research because practically all patients with this type of diagnosis have trigger points in these muscles, and dry needling technique is one of the best for its treatment, but has the disadvantage that it produces post dry needling pain of 48 hours and there is not enough information, or consensus on which method is better to reduce post dry needling pain. This study aims to prove wich technique is most useful in reducing pain post dry needling for the treatment of trigger points in the triceps sural muscle in ankle post fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 60 years of age.
* Man or woman.
* At least one trigger point, active or latent, in the triceps sural muscle of the fractured ankle.
* Perform full load without using technical aids.

Exclusion Criteria:

* Use of analgesics.
* Insurmountable fear of needles.
* Immune disease.
* Clotting disorders.
* Sensory disorders.
* Psychiatric / psychological illness.
* Cancer.
* Rheumatic diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived pain intensity | Change from baseline (baseline and immediately after treatment)
  Pain will be measured by the Visual Analog Scale for pain (VAS) from 0 to 10, where higher values represent a worse outcome.
Ankle Range of Motion (ROM) | Change from baseline (baseline and immediately after treatment)
  It is the degree of angular movement allowed by the ankle joint measured by kinovea.

SECONDARY OUTCOMES:
Muscular strength of triceps sural | Change from baseline (baseline and immediately after treatment)
  By means of the heel rise test, the patient must perform a bipodal plantiflexion measured in the maximum number of repetitions in 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario San Jose, Santiago, Chile